CLINICAL TRIAL: NCT05370560
Title: Plasma Transthyretin Levels and Risk of Type 2 Diabetes Mellitus and Impaired Glucose Regulation in a Chinese Population
Brief Title: Plasma Transthyretin Levels and Risk of Type 2 Diabetes Mellitus and Impaired Glucose Regulation
Status: Completed | Type: Observational
Sponsor: Liegang Liu (Other)
Responsible Party: Sponsor-Investigator, Liegang Liu, Professor, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Other Study IDs: YR202205
Record Dates: First submitted 2022-05-07; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes; Impaired Glucose Regulation
Keywords: transthyretin; type 2 diabetes; impaired glucose regulation
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Type 2 diabetes mellitus: In this case-control study, T2DM was diagnosed according to the diagnostic criteria recommended by the WHO in 1999. T2DM was confirmed when fasting plasma glucose (FPG) ≥ 7.0 mmol/L and/or 2-h post-glucose load (OGTT2h) ≥ 11.1 mmol/L.
  Interventions: Other: Plasma transthyretin concentration
- Impaired glucose regulation: In this case-control study, IGR was diagnosed according to the diagnostic criteria recommended by the WHO in 1999. IGR was defined as impaired fasting glucose ([FPG] ≥ 6.1 mmol/L and < 7.0 mmol/L, and [OGTT2h] < 7.8 mmol/L) and/or impaired glucose tolerance (FPG < 7.0 mmol/L, and OGTT2h ≥ 7.8 mmol/L and < 11.1 mmol/L).
  Interventions: Other: Plasma transthyretin concentration
- Control: Those with FPG < 6.1 mmol/L and OGTT2h < 7.8 mmol/L were considered controls.
  Interventions: Other: Plasma transthyretin concentration

INTERVENTIONS:
Other: Plasma transthyretin concentration — Plasma transthyretin concentrations were measured by BS 200 Autoanalyser (Mindray, Shenzhen, China) using immunoturbidimetric method.

SUMMARY:
Objective: To investigate the association between plasma transthyretin levels and risk of newly diagnosed type 2 diabetes mellitus (T2DM) and impaired glucose regulation (IGR) in a Chinese population.

Design: We performed a case-control study, including 1,244 newly diagnosed T2DM patients, 837 newly diagnosed IGR patients, and 1,244 individuals with normal glucose tolerance (NGT). The diagnostic criteria were recommended by World Health Organization in 1999. All cases were recruited from patients who, for the first time, received a diagnosis of T2DM in the Department of Endocrinology, Tongji Hospital, Tongji Medical College, Wuhan, China, from December 2010 to December 2016. Concomitantly, general population undergoing a routine health checkup in the same hospital were enrolled as controls. The inclusion criteria were age ≥ 30 years, BMI < 40 kg/m2, and no history of diagnosis of diabetes or receiving pharmacological treatment for hypertension and hyperlipidemia. Participants with clinically significant neurological, endocrinological, psychological or other systemic diseases, as well as acute illness or chronic inflammatory or infectious diseases, were excluded from the present study. Written informed consent was obtained from each participant. Besides, cases were stringently matched to controls in a 1:1 ratio, based on sex and age (± 3 years). All participants enrolled were of Han ethnicity, and gave a commitment of taking no medication known affecting glucose tolerance or insulin secretion before participating in the study. Fasting blood samples were collected in EDTA-anticoagulative tubes and separated for plasma within 1 h. Then plasma was kept at -80℃ prior to analyses. Plasma transthyretin levels were measured by BS 200 Autoanalyser (Mindray, Shenzhen, China) using immunoturbidimetric method.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 30 years, BMI < 40 kg/m2, and no history of diagnosis of diabetes or receiving pharmacological treatment for hypertension and hyperlipidemia

Exclusion Criteria:

* Clinically significant neurological, endocrinological, psychological or other systemic diseases, as well as acute illness or chronic inflammatory or infectious diseases.

Incomplete basic information.

Ages: 24 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All the participants enrolled were of Chinese Han ethnicity. They gave informed written consent to the study and did not take any medication known to affect glucose tolerance or insulin secretion before participation.
Sampling Method: Probability Sample
Enrollment: 3325 (Actual)
Dates: Start 2010-12-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Type 2 diabetes mellitus | From December 2010 to December 2016
  In the case-control study, type 2 diabetes mellitus was diagnosed in accordance with the diagnostic criteria recommended by WHO in 1999.